CLINICAL TRIAL: NCT05317637
Title: Cardiopulmonary Outcomes in Osteogenesis Imperfecta: BBD7708
Status: Active, not recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Brendan Lee, Consortium PI, Baylor College of Medicine
Other Study IDs: H49848
Record Dates: First submitted 2021-08-23; First posted 2022-04-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2024-12

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with OI: 18 participants will be enrolled through in this pilot study. Interested males with OI will be preferred over females to compensate for our highly female original cohort and determine if sexual dimorphism exists for cardiopulmonary outcomes in people with OI.
  This study is cross-sectional. At the participant's one study visit, data will be obtained at a single point in time and reflect the patients' current condition. All efforts will be made to complete all data collection and testing on the same day. However, procedures completed within ±12 months will be accepted. Evaluations will include family and medical history, self-report questionnaires, physical evaluation, diagnostic studies, and radiographic studies. Participants will be enrolled regardless of OI type since BWT, a finding we are attempting to validate, was observed in all types of OI. Smokers will not be excluded.

SUMMARY:
Osteogenesis imperfecta (OI) is a group of congenital and heritable bone disorders that currently affects at least 50,000 people in the United States. OI varies in severity from perinatally lethal to mild forms. The majority of cases is caused by a dominant mutation in type I collagen genes (COL1α1 and COL1α2), altering the quantity or quality of type I collagen.

Although OI is typically characterized as a disease of the bone, it is perhaps more accurately described as a connective tissue disorder. Type I collagen is a major constituent of lung connective tissue. Respiratory insufficiency is the leading cause of death in patients with OI. Thus, it is important and necessary to understand the etiology of the restrictive pulmonary physiology in the OI population.

DETAILED DESCRIPTION:
This study is cross-sectional. At the participant's one study visit, data will be obtained at a single point in time and reflect the patients' current condition. Evaluations will include family and medical history, self-report questionnaires, physical evaluation, diagnostic studies, and radiographic studies. Eighteen participants will be enrolled, ideally within one year. Participants will be enrolled regardless of OI type since Bronchial Wall Thickening, a finding we are attempting to validate, was observed in all types of OI. Interested males with OI will be preferred over females to compensate for our highly female original cohort and determine if sexual dimorphism exists for cardiopulmonary outcomes in people with OI. Smokers will not be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are able to give informed consent or have a legally authorized representative capable of giving consent on the subject's behalf
* Individuals ages 18 and older of all races and sexes
* Individuals who have been diagnosed with OI clinically and/or genetically

Exclusion Criteria:

* Individuals diagnosed with respiratory illness within 6 weeks of enrollment or undergoing diagnostic studies for an active illness.
* Individuals with other skeletal dysplasia or genetic diagnosis
* Individuals diagnosed with cardiopulmonary comorbidities that affect lung compliance

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals with Osteogenesis Imperfecta
Sampling Method: Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
proportion of restrictive lung physiology | 12 months
  FEV1/FVC greater than or equal to 80%, which is obtained from PFT

SECONDARY OUTCOMES:
Presence and severity of Bronchial Wall Thickening | 12 months
  measurement of percent of bronchial diameter subsumed by wall thickness
Vital lung capacity | 12 months
  Vital capacity/total lung capacity/chest volume prediction based on 1) readings by trained chest CT readers and 2) 3-D lung imaging calculation
Presences of pulmonary fibrosis | 12 months
  Presence of pulmonary fibrosis based on readings by trained chest CT readers
Change in lung tissue | 12 months
  location of bronchiectasis, and presence of atelectasis based on readings by trained chest CT readers

OTHER OUTCOMES:
Scoliosis | 12 months
  Measurement of spinal scoliosis, kyphosis, lordosis and vertebral fractures including curve measurement based on standing plane films of thorax/abdomen exposed for bone imaging

CONTACTS AND LOCATIONS:
Overall Officials: Vernon Sutton, MD, Principal Investigator — Baylor College of Medicine; Kathleen Raggio, Study Chair — Hospital for Special Surgery, New York
Locations (3):
- United States (3):
  - University of California Los Angeles, Los Angeles, California
  - Kennedy Krieger Institute / Hugo W. Moser Research Institute, Baltimore, Maryland
  - Hospital for Special Surgery, New York, New York

IPD SHARING:
Plan to Share IPD: No